CLINICAL TRIAL: NCT02468739
Title: The Effect of Monosialotetrahexosyl Ganglioside (GM1) in Prevention of Taxanes Induced Neurotoxicity in Breast Cancer Patients Who Received Taxanes-based Adjuvant Chemotherapy: A Multi-center, Randomized, Placebo-controlled Trial
Brief Title: Effect of GM1 in Prevention of Taxanes Induced Neurotoxicity in Operable Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYSUCC-013
Record Dates: First submitted 2015-05-14; First posted 2015-06-11 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganglioside-monosialic acid arm (Experimental): Patients will receive treatment of adjuvant chemotherapy. Ganglioside-monosialic acid(GM1, 80mg per day) will be given at 1 day before the start of chemotherapy for three days (Day -1, 1 and 2).
  Chemotherapy regimens:
  Epirubicin (90 mg/m2) combined with cyclophosphamide (600 mg/m2) followed by paclitaxel (175 mg/m2 *4 cycles) after four courses of chemotherapy; Epirubicin (90 mg/m2) combined with cyclophosphamide (600 mg/m2) followed by docetaxel (75 mg/m2 *4 cycles) after four course of chemotherapy; Docetaxel (75 mg/m2 q21d) combined with cyclophosphamide (600 mg/m2) for four courses.
  The first day (D1) of each cycle is treated with taxane-based chemotherapy. 14-21 days are usually as one cycle. The methods of pretreatment and hydration shall be decided by the physicians.
  Interventions: Drug: Ganglioside-monosialic acid
- placebo arm (Placebo Comparator): Patients will receive treatment of adjuvant chemotherapy. Placebo will be given at 1 day before the start of chemotherapy for three days (Day -1, 1 and 2).
  Chemotherapy regimens:
  Epirubicin (90 mg/m2) combined with cyclophosphamide (600 mg/m2) followed by paclitaxel (175 mg/m2 *4 cycles) after four courses of chemotherapy; Epirubicin (90 mg/m2) combined with cyclophosphamide (600 mg/m2) followed by docetaxel (75 mg/m2 *4 cycles) after four course of chemotherapy; Docetaxel (75 mg/m2 q21d) combined with cyclophosphamide (600 mg/m2) for four courses.
  The first day (D1) of each cycle is treated with taxane-based chemotherapy. 14-21 days are usually as one cycle. The methods of pretreatment and hydration shall be decided by the physicians.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ganglioside-monosialic acid — Ganglioside-monosialic sodium is added into to 250 ml of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 3 days. The first dose is given at 1 day before the start of the chemotherapy.(day -1, day 1 and day2). The dosages of GM1 are 80mg per day.
  Other Names: GM1
  Arms: Ganglioside-monosialic acid arm
Drug: placebo — Placebo is added into to 250 ml of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 3 days. The first dose is given at 1 day before the start of the chemotherapy.(day -1, day 1 and day2).
  Arms: placebo arm

SUMMARY:
Background: Taxane plays a key role in the treatment of breast cancer and taxane-induced peripheral neuropathy (TIPN) is a dose-limiting adverse effect leading to treatment discontinuation. Ganglioside-monosialic acid (GM1) functions as a neuroprotective factor. However, the effects of GM1 on TIPN in breast cancer patients remains unknown.

Purpose: This randomized phase III trial is designed to evaluate the potential effects of GM1 for preventing TIPN in breast cancer patients.

DETAILED DESCRIPTION:
Introduction： Taxanes is a key agent in the treatment of breast cancer. However, peripheral neuropathy markedly limits the use of taxanes. Unfortunately, current studies have neither revealed a clear mechanism nor established an effective treatment for Taxane-induced peripheral neuropathy (TIPN). Monosialotetrahexosyl ganglioside (GM1) functions as a neuroprotective factor. This multi-center, randomized, placebo-controlled trial was performed to assess the efficacy of GM1 fo preventing taxanes induced neurotoxicity in operable breast cancer patients who received taxanes-based adjuvant chemotherapy.

OBJECTIVES:

Primary Objective:

To evaluate the efficacy of gangliosides in the prevention of neurotoxicity in breast cancer patients treated with taxane-based chemotherapy. That is, to compare the differences in the scores of Functional Assessment of Cancer Treatment Neurotoxicity (FACT-Ntx) between the patients treated by GM1(the treatment group) and the placebo (the control group) at 2 weeks after completion of 4-cycles of taxane-based chemotherapy.

Secondary

* To compare the differences in the scores of Eastern Cooperative Oncology Group neuropathy scale between the patients treated by gangliosides (the experimental group) and the placebo (the control group);
* Tocompare the incidence of neurotoxic adverse events caused by taxane-based chemotherapy. That is, the difference between the patients of chemotherapy treated by gangliosides (the experimental group) and the placebo (the control group) in terms of the incidence of neurotoxicity (graded according to the NCI-CTCAE version 4.0 grading scale);
* Assess the safety and tolerance of the two treatment groups (ganglioside and placebo groups).

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients with early-stage breast cancer planning to receive taxane-based adjuvant chemotherapy were randomly assigned to receive GM1 (80 mg, Day -1 to Day 2) or placebo treatment.

Treatment group: Monosialotetrahexosylganglioside sodium is added into 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 3 days. The first dose is given at 1 day before the start of the chemotherapy. At the same time, the patients are treated with a taxane-based chemotherapy selected by the investigators.

Placebo group: Placebo is added into 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 3 days. The first dose is given at 1 day before the start of the chemotherapy. At the same time, the patients are treated with a taxane-based chemotherapy selected by the investigators.

The screening and baseline peripheral neurotoxicity assessment was performed 1 day before the start of the first course of taxane-containing chemotherapy.

The subjects will be treated by the study drugs according to the schedule until the completion of established taxane-based adjuvant chemotherapy, the onset of unacceptable toxicity, or when the patient withdraw from the study voluntarily.

Endpoint assessments including FACT-Ntx subscale, CTCAE version 4.0 grading scale and ENS subscales were performed at 2 weeks after each course of chemotherapy. Additional long-term assessments were performed at 3 months, 6 months and 1 year after the end of chemotherapy. The follow-up will be carried out until 2 years after the enrollment time of the last patient.

ELIGIBILITY:
Enrollment Criteria:

* Female patients with histologically confirmed early-stage breast cancer at the age of ≥18 and ≤75 , who have received radical surgical treatment of breast cancer (including modified radical mastectomy and breast-conserving surgery) while have not received neoadjuvant chemotherapy. EC*4-T*4 chemotherapy (T is paclitaxel or docetaxel) protocol is expected, and there is no herceptin indication or the patients are voluntarily not to be treated with herceptin.
* Patients with KPS（Karnofsky Performance Status) scores ≥ 80;
* Patients with ECOG score ≤ 1;
* Expected survival ≥ 3 months;
* The functional level of main organs must meet the following requirements (no blood transfusion, no leucocyte or platelet-ascending drugs used within 2 weeks before screening):1)Blood Routine: Neutrophil (ANC) ≥ 1.5 x 109/L;Platelets (PLT) ≥ 90 x 109/L; Hemoglobin (Hb) ≥ 90 g/L;2) Blood Biochemistry Total bilirubin (TBIL) ≤ 1.5 x ULN;L-Alanine (ALT) and aspartic transaminase (AST) ≤ 2 x ULN;Blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 x ULN;
* Cooperate to complete questionnaire accurately recording occurrence and severity of neurotoxicity
* Sign the informed consent form.

Exclusion Criteria:

* There are any toxicity events of peripheral nervous system before enrollment, including: FACT-Ntx subscale score < 44;≥ Grade 1 peripheral toxicity according to CTCAE Version 4.0 rating scale;≥ Grade 1 peripheral toxicity according to ENS rating scale;All other pathological symptoms or diseases might affect the evaluation of adverse neurotoxic effects
* Patients having received other drug treatments might cause similar adverse neurotoxic effects within 4 weeks prior to the treatment of this protocol, or receive concurrent neurotoxic drugs. Including: Taxanes or analogues; Vinca alkaloids or analogues; Platinums or analogues; Cytarabine, thalidomide, bortezomib, or procarbazine; Other drugs or treatments might cause peripheral neurotoxicity
* Patients in poor general conditions, with KPS (Karnofsky performance status) scores < 80;
* Pregnant or lactating women；
* Patients (female) having the possibility of fertility but unwilling or not taking effective contraceptive measures
* Patients also having other neurological abnormalities who cannot accurately record the occurrence and severity of neurotoxicity;
* Patients known allergy to trial drugs or excipient compositions of these products;
* Patients with inherited glucose and lipid metabolism abnormalities (gangliosidosis such as amaurotic family idiocy and retinopathy);
* Patients not suitable for treatment of ganglioside;
* Active infection (depending on the judgment of investigators);
* Patients with serious concurrent diseases might harmful to safety and interfere the scheduled treatment or concomitant diseases might affect the completion of the study, depending on the judgment of investigators.
* Patients with a history of definite neurological or dysphrenia, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the Functional Assessment of Cancer Treatment Neurotoxicity (FACT-Ntx) subscale between groups at 2 weeks after the 4-cycle chemotherapy | Day 1 of Week 1 to 1 year after the last course of chemotherapy
  The primary endpoint was assessed using the Functional Assessment of Cancer Treatment, Gynecologic Oncology Group Neurotoxicity (FACT -Ntx) subscale at 2 weeks after completion of 4-cycles of taxane-based chemotherapy.
  FACT-Ntx subscales contains 11 items including numbness, tingling, and discomfort in the hands or feet; difficulty hearing or tinnitus; joint pain or muscle cramps; weakness or fatigue; or trouble walking, buttoning buttons, or feeling small shapes when placed in the hand; feeling pain or hard to breath when exposed to low temperature. Each Items is scored from 0 to 4 with a total score of 44; higher scores indicate better performance.
  A 5-point difference in the FACT-Ntx subscale scores between groups is considered clinically meaningful.
  The FACT-Ntx subscales assessments were performed at 2 weeks after each course of chemotherapy. Additional long-term assessments were performed at 3 months, 6 months and 1 year after the end of chemotherapy.

SECONDARY OUTCOMES:
neurotoxicity evaluated by NCI-CTCAE version 4.0 grading scale | 1 monthDay 1 of Week 1 to 1 year after the last course of chemotherapy
  neurotoxicity evaluated by NCI-CTCAE version 4.0 grading scale which classified symptoms as grade 0, 1, 2, 3, or 4. Higher scores indicate more severe neurotoxicity.
  The NCI-CTCAE version 4.0 assessments were performed at 2 weeks after each course of chemotherapy. Additional long-term assessments were performed at 3 months, 6 months and 1 year after the end of chemotherapy.
neurotoxicity evaluated by the Eastern Cooperative Oncology Group neuropathy scale (ENS) subscales of sensory neuropathy, motor neurotoxicity, and neurogenic constipation. | Day 1 of Week 1 to 1 year after the last course of chemotherapy
  The ENS subscales (from 0 to 4 scale) of sensory neuropathy, motor neurotoxicity, and neurogenic constipation were examined. For each of these scales, lower scores indicate better performance.
  The ENS subscales assessments were performed at 2 weeks after each course of chemotherapy. Additional long-term assessments were performed at 3 months, 6 months and 1 year after the end of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Yuan, M.D., Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No